CLINICAL TRIAL: NCT02263118
Title: A Mobile-health Pilot Experiment Targeting Mothers With Newborns in Rural Areas of San Juan Sacatepequez, Guatemala, in the Context of Exclusive Breastfeeding Practices
Brief Title: A Mobile-health Pilot Experiment Targeting Mothers With Newborns in Rural Areas of San Juan Sacatepequez, Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco Marroquín (Other)
Collaborators: Ecole Polytechnique, France (Unknown); The SHM Foundation, UK (Unknown)
Responsible Party: Principal Investigator, José Tomás PRIETO, PhD, Dr. Jose Tomas Prieto, Universidad Francisco Marroquín
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CE/FM UFM 0062-13
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Exclusive Breastfeeding; Co-production of Health in Communities
Keywords: breastfeeding; rural; m-health; mHealth; Patojitos; Guatemala; exclusive breastfeeding; mobile; eHealth; e-health
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- Uni-directional SMS (Experimental): Participants in this group received breastfeeding promoting messages based on the MAMA (http://www.mobilemamaalliance.org/) breastfeeding database. Individuals could only receive text messages.
  Interventions: Other: Uni-directional SMS; Device: Feature phone
- Virtual communities (Experimental): Participants were made part of virtual communities in which could exchange about infant's health as groups, via SMS, following the SHM Foundation's (http://www.shmfoundation.org/) m-health methodology.
  Interventions: Other: Uni-directional SMS; Device: Feature phone; Other: Virtual communities
- Hybrid setup (Experimental): Participants were made part of virtual communities in which they could exchange about infant's health as groups, via SMS. Additionally, a health professional was included in the virtual community.
  Interventions: Other: Uni-directional SMS; Device: Feature phone; Other: Virtual communities; Other: Hybrid setup
- Control group (Experimental): Individuals were given a feature phone (simple mobile phone)
  Interventions: Device: Feature phone

INTERVENTIONS:
Other: Uni-directional SMS — Exposure to breastfeeding promoting SMSs
  Arms: Hybrid setup; Uni-directional SMS; Virtual communities
Device: Feature phone — Participants were given a feature phone.
Other: Virtual communities — Exposure to virtual community communication via SMS
  Arms: Hybrid setup; Virtual communities
Other: Hybrid setup — Exposure to virtual community and access to communications with health professional via SMS
  Arms: Hybrid setup

SUMMARY:
The purpose of this study was to determine whether exposure to m-health platforms promoting recommended breastfeeding practices was effective in transmitting the exclusive breastfeeding message to participant mothers, and in improving weight evolution of infants.

ELIGIBILITY:
Inclusion Criteria:

* Can read
* Has a baby of less than 4 months of age OR is in her 8th month of pregnancy

Exclusion Criteria:

* Cannot read
* Does not have a newborn

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Tulio Rodriguez, MD, Study Chair — Universidad Francisco Marroquin, Guatemala; Jose Tomas Prieto, Principal Investigator — Ecole Polytechnique, France; Universidad Francisco Marroquin, Guatemala

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group
Started | 24 | 32 | 30 | 14
Completed | 20 | 24 | 22 | 12
Not Completed | 4 | 8 | 8 | 2

BASELINE CHARACTERISTICS:
Population: Indigenous women from San Juan Sacatepequez
Groups:
- Total: Total of all reporting groups
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group | Total
Number analyzed (Participants) | 20 | 24 | 22 | 12 | 78
Age, Customized [Number; unit: participants]
  16-22 years | 9 | 11 | 10 | 2 | 32
  23-30 years | 9 | 10 | 9 | 7 | 35
  >30 years | 2 | 3 | 3 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participant's baby
  Participants
    Female | 12 | 14 | 5 | 6 | 37
    Male | 8 | 10 | 17 | 6 | 41
Maternal experience [Number; unit: participants] — Does the participant have other children?
  participants
    Yes | 11 | 12 | 13 | 8 | 44
    No | 9 | 12 | 9 | 4 | 34
Education [Number; unit: participants] — Women's education
  participants
    None | 2 | 3 | 1 | 1 | 7
    Some primary school education | 16 | 18 | 18 | 7 | 59
    Some high school education | 2 | 3 | 3 | 3 | 11
    > High school | 0 | 0 | 0 | 1 | 1
Aware of exclusive breastfeeding message [Number; unit: participants] — Was the participant aware of exclusive breastfeeding practice at enrollment?
  participants
    Aware | 8 | 18 | 10 | 9 | 45
    Not Aware | 12 | 6 | 12 | 3 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Knowledge
Description: Specifically, we were interested in: the number of participants who switched from an incorrect to a correct knowledge regarding exclusive breastfeeding during the experiment (learned the message); the number of participants who had a correct knowledge but switched to an incorrect one during the experiment (forgot the message); the number of participants who had an incorrect knowledge and kept it until the end of the experiment (continued to be unaware); the number of participants who had a correct knowledge and kept it until the end of the experiment (remembered the message).
Time Frame: December 2013 - May 2014, 23 weeks
Measure: Number; unit: participants
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group
Number analyzed (Participants) | 20 | 24 | 22 | 12
participants
  Learned it | 12 | 2 | 11 | 3
  Forgot it | 0 | 8 | 0 | 4
  Remembered it | 8 | 10 | 10 | 5
  Continued to be unaware at the end of experiment | 0 | 4 | 1 | 0

2. Secondary Outcome: Qualitative Nature of Health-related Text-messages
Description: Specifically, we were interested in classifying individual text-messages as social support or health related.
Time Frame: December 2013 - May 2014, 23 weeks
Measure: Number; unit: Number of text messages
Units Other Than Participants: Text messages shared in groups
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group
Number analyzed (Participants) | 0 | 24 | 22 | 0
Number analyzed (Text messages shared in groups) | 0 | 2793 | 909 | 0
Number of text messages
  Health related messages |  | 761 | 501 |
  Social support related messages |  | 1961 | 356 |
  Other messages |  | 71 | 52 |

3. Secondary Outcome: Number of Text-messages Exchanged in Virtual Communities
Description: We were interested in the activity of virtual communities in terms of sent text-messages.
Time Frame: December 2013 - May 2014, 23 weeks
Population: In "virtual communities", participants were added to 1 of 3 peer-to-peer groups. They could communicate by sending SMSs to a short-code number. In the "hybrid setup", participants were added to 1 of 3 peer-to-peer groups, but in addition received information regarding breastfeeding practices and could communicate with a health professional.
Measure: Number; unit: Number of text messages
Groups:
- Uni-directional SMS: There were no virtual communities in this group: participants in this group received breastfeeding promoting messages based on the MAMA (http://www.mobilemamaalliance.org/) breastfeeding database. Individuals could only receive text messages.
  Uni-directional SMS: Exposure to breastfeeding promoting SMSs
  Feature phone: Participants were given a feature phone.
- Control Group: There were no virtual communities in this group: individuals were given a feature phone (simple mobile phone)
  Feature phone: Participants were given a feature phone.
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group
Number analyzed (Participants) | 0 | 24 | 22 | 0
Number of text messages |  | 2793 | 909 |

4. Secondary Outcome: Mean Change in Weight-for-Age Z-score
Description: We used the World Health Organization Anthro software (http://www.who.int/childgrowth/software/en/) to calculate z-scores for the weight-for-age anthropometric indicator of participants' infants at the beginning and at the end of the project. The software is based on the WHO Child Growth Standards and allowed to compare measurements of infants to the normal growth standards. The Z-score indicates the number of standard deviations away from the mean. The indicator is particularly useful to detect abnormal growth patterns in infants' development. For instance, an infant whose weight falls in the -2 z-score for the weight-for-age anthropometric indicator is underweight. Below -3, the child is severely underweight. Similarly, a child whose weight-for-age is above a +1 z-score may have a growth problem.
  We report the mean change of the z-scores for the weight-for-age anthropomorphic indicator of participants' babies.
Time Frame: Baseline at December 2013 and 23 weeks later in May 2014
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group
Number analyzed (Participants) | 20 | 24 | 22 | 12
z-score | -0.064 [-0.355 to 0.228] | 0.030 [-0.282 to 0.343] | 0.199 [-0.331 to 0.728] | -0.197 [-0.834 to 0.441]

ADVERSE EVENTS:
Time Frame: 23 weeks
Arm/Group | Uni-directional SMS | Virtual Communities | Hybrid Setup | Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24 | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 0/20 | 0/24 | 0/22 | 0/12

LIMITATIONS AND CAVEATS:
Future work could consider a wider time span and inspect complementary instruments to ensure consistency between answers to interviews and behaviour. SMSs in virtual communities could be further analyzed to locate longitudinal changes in knowledge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No